CLINICAL TRIAL: NCT03062098
Title: Optimizing the Technique of Embryo Transfer in IVF Using Better Imaging Guidance
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Primary investigator retired, rest of staff cannot continue
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 0229-16-RMB
Record Dates: First submitted 2017-02-13; First posted 2017-02-23 (Actual); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Fertilization in Vitro
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IVF patients (Experimental): IVF patients before embryo transfer. Before performing embryo transfer in the routine manner, ten patients will be asked to participate in the study. After signing informed consent, participants will undergo the experimental procedure: Speculum will be placed to visualize the cervix. The thin ultrasound probe will be places posterior to the cervix. While viewing the image on the ultrasound screen, the probe will be moved manually to obtain the best imaging of the cervical canal. An empty embryo transfer catheter will be introduced to the cervical canal and will be advanced under ultrasound imaging up to the internal os. The catheter will be withdrawn, and routine embryo transfer will follow.
  Interventions: Device: ultrasound imaging

INTERVENTIONS:
Device: ultrasound imaging — Ultrasound imaging during embryo transfer using a small vaginal probe.

SUMMARY:
This trial seeks to improve ultrasound imaging during embryo transfer in IVF by using a small, high resolution ultrasound probe used routinely for cardiac imaging in children.

DETAILED DESCRIPTION:
Since the first pregnancy using IVF was achieved nearly 40 years ago, many aspects of this procedure have undergone significant progress. In contrast, the technique of embryo transfer (ET) has remained relatively unchanged. A simple yet critical element in the final step of IVF, ET has received little attention. In general, the procedure starts by placing a speculum in the vagina to visualize the cervix, which is cleansed with saline solution or culture media. A transfer catheter is loaded with the embryos is inserted through the cervical canal and advanced into the uterine cavity where the embryos are deposited.

The catheter is then withdrawn and handed to the embryologist, who inspects it for retained embryos. Ultrasound (US) guidance is used to facilitate atraumatic insertion of the catheter, as well as ensure correct location in the uterine cavity.

The available evidence suggests that there is a benefit of using US guidance during ET (Teixeira et al, Ultrasound Obstet Gynecol. 201;45:139-48, Abou-Setta et al, Fertil Steril. 2007;88:333-41).

High quality US imaging is difficult to achieve if the distance from the abdominal wall to the uterus is big (thick abdominal wall, retro-verted uterus), or if the bladder is not full enough.

High resolution US imaging dictates short distance between the US transducer and the organ of interest (in our case cervical canal and endometrium). Previous effort in that direction was done using a vaginal US probe. However, this instrumentation makes the ET technique cumbersome and difficult to perform. We hypothesize that a significant advantage in imaging quality can be achieved by placing a flat or concave high frequency US transducer in the posterior fornix as an extension of the posterior speculum blade.

Our overarching goal is to develop new ET procedure; this procedure will be dependent on precise and high resolution imaging. For that goal we consulted with ultrasound experts that recommended the use of dedicated probe. After a thorough review we found a probe (Philips 21381A / T6207) that is used for pediatric transesophageal applications with operating frequency of 4-7 Megahetz.

As part of the embryo transfer, the investigators plan to insert the above probe into the posterior fornix. The investigators will then evaluate the visualization abilities of placing a probe closer to the uterus. The aim is to define the ultrasound image parameters for ET. The information will be used to define the technical specification for a "tailor made" ET probe.

ELIGIBILITY:
Inclusion Criteria: IVF patients before embryo transfer. -

Exclusion Criteria: IVF patients not willing to participate

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — IVF patients - all females
Enrollment: 0 (Actual)
Dates: Start 2017-05-15 (Estimated); Primary Completion 2017-07-01 (Estimated); Study Completion 2017-09-01 (Estimated)

PRIMARY OUTCOMES:
Imaging quality | About 1 minute
  Characterization of exact ultrasound image planes while placing an ultrasound probe within the posterior fornix, for anatomical optimization

CONTACTS AND LOCATIONS:
Locations (1):
- IVF Unit, Rambam medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No